CLINICAL TRIAL: NCT07015658
Title: Clinical Effects of Moxibustion Combined With Tailored Baduanjin Exercise Programs on Early Postoperative Rehabilitation in Lumbar Disc Herniation Patients Undergoing Minimally Invasive Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suyun Liu (Other)
Responsible Party: Sponsor-Investigator, Suyun Liu, Suyun Liu, Second Affiliated Hospital of Nanchang University
Organization: Second Affiliated Hospital of Nanchang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIT-I-2025-062
Record Dates: First submitted 2025-06-04; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Lumbar Disc Herniations
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Moxibustion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): 1. Routine nursing measures: Postoperatively, routine basic treatments such as preventing infection, anti-inflammatory and analgesic therapy, nourishing the nerves, eliminating edema, and suppressing acid and protecting the stomach are provided. After discharge, patients are instructed to take anti-inflammatory and analgesic drugs and nourishing nerve drugs as prescribed. Systematic nursing interventions are carried out after the operation, including psychological intervention and health education; avoid prolonged sitting, prolonged standing, heavy lifting and physical labor. Adopt the correct standing and walking postures, and use a waist brace for protected bed mobility for one month. After discharge, instruct patients to visit the clinic for regular follow-ups and consult as needed.
  Interventions: Procedure: Conventional intervention
- Baduanjin Group (Experimental): The Baduanjin protocol, based on China's 2003 General Administration of Sport standard, was modified by professional physiotherapists for targeted adaptations, with nurses receiving specialized training. Patients viewed step-by-step instructional clips upon admission alongside a full-length routine video. Standard postoperative rehabilitation was maintained during Weeks 1-2. At Week 3, patients demonstrating adequate wound healing and unimpaired static lumbar muscle contraction performed Baduanjin exercises wearing a lumbar brace, supervised by trained nurses for movement correction. The brace was discontinued after 8 weeks. Modified professional videos with background music were distributed via WeChat/official accounts twice daily (30min/session, 5 days/week) for 13 weeks (total ≥2000min). Duration/frequency adjustments were permitted based on individual recovery and physician recommendations post-intervention.
  Interventions: Procedure: Baduanjin; Procedure: Conventional intervention
- Combined Intervention Group (Experimental): Moxibustion was performed at acupoints including Yaoyangguan (GV3), Shenshu (BL23), Dachangshu (BL25, affected side), Chengfu (BL36), Mingmen (GV4), Weizhong (BL40, affected side), Taixi (KI3), Fuliu (KI7), Zhishi (BL52), Zusanli (ST36), and Ashi points. Using five-year-aged Qizhou mugwort, the patient's treatment areas were fully exposed in a comfortable position. The moxa stick was held 3-4 cm from the skin with intensity adjusted to patient tolerance to prevent burns. The circular moxibustion technique was applied for 3-5 minutes per acupoint until the skin exhibited erythema, perspiration, or mottling, or until the patient experienced warmth, distension, itchiness, or perceived moxa-heat propagation. Treatment commenced at postoperative Week 3 following evaluation of satisfactory wound healing, administered three times weekly for four consecutive weeks.
  Interventions: Procedure: Baduanjin; Procedure: Moxibustion; Procedure: Conventional intervention

INTERVENTIONS:
Procedure: Baduanjin — The Baduanjin protocol, based on China's 2003 General Administration of Sport standard, was modified by professional physiotherapists for targeted adaptations, with nurses receiving specialized training. Patients viewed step-by-step instructional clips upon admission alongside a full-length routine video. Standard postoperative rehabilitation was maintained during Weeks 1-2. At Week 3, patients demonstrating adequate wound healing and unimpaired static lumbar muscle contraction performed Baduanjin exercises wearing a lumbar brace, supervised by trained nurses for movement correction. The brace was discontinued after 8 weeks. Modified professional videos with background music were distributed via WeChat/official accounts twice daily (30min/session, 5 days/week) for 13 weeks (total ≥2000min). Duration/frequency adjustments were permitted based on individual recovery and physician recommendations post-intervention.
  Arms: Baduanjin Group; Combined Intervention Group
Procedure: Moxibustion — Moxibustion was performed at acupoints including Yaoyangguan (GV3), Shenshu (BL23), Dachangshu (BL25, affected side), Chengfu (BL36), Mingmen (GV4), Weizhong (BL40, affected side), Taixi (KI3), Fuliu (KI7), Zhishi (BL52), Zusanli (ST36), and Ashi points. Using five-year-aged Qizhou mugwort, the patient's treatment areas were fully exposed in a comfortable position. The moxa stick was held 3-4 cm from the skin with intensity adjusted to patient tolerance to prevent burns. The circular moxibustion technique was applied for 3-5 minutes per acupoint until the skin exhibited erythema, perspiration, or mottling, or until the patient experienced warmth, distension, itchiness, or perceived moxa-heat propagation. Treatment commenced at postoperative Week 3 following evaluation of satisfactory wound healing, administered three times weekly for four consecutive weeks.
  Arms: Combined Intervention Group
Procedure: Conventional intervention — Postoperative Rehabilitation Exercises: Week 1: Ankle Pump Exercises: Start after anesthesia. Slowly rotate/invert, dorsiflex/plantarflex ankles. Hold each position 10-15s. 30 min/set, 6 sets/day, until ambulation. Straight Leg Raising (SLR): Start Day 2, supine. Elevate leg >30°. Progress from passive to active hold. Hold 5-10s/rep, 10-20 reps/set. 3 sets (morning/noon/night) daily for 15 days. Week 2: Supine hip/knee flexion exercises in bed. Hold each flexion 3-5s. 30-50 reps/set. 2 sets/day. Weeks 3-4: Start back muscle training (e.g., bridge/bird-dog poses). Months 1-3: Gradually increase back exercise frequency/difficulty. Perform flexion, extension, lateral flexion, and rotation wearing a lumbar brace. Intensity/reps based on tolerance.

SUMMARY:
This study is a single-center randomized controlled trial, aiming to explore the effect of moxibustion combined with the modified Baduanjin exercise regimen on the early rehabilitation of patients with lumbar disc herniation (LDH) after minimally invasive surgery. A total of 120 patients were included in the study and randomly divided into the control group (conventional treatment and rehabilitation care), the Baduanjin group (conventional treatment + modified Baduanjin), and the combined intervention group (conventional treatment + Baduanjin + moxibustion). By comparing the visual pain scores (VAS), lumbar function scores (JOA), lumbar range of motion, and anxiety scale (HAMA) changes at 1 day, 1 month, and 3 months after surgery, the study evaluated the improvement effect of the integrated traditional Chinese medicine and Western medicine rehabilitation plan on postoperative pain relief, functional recovery, and psychological state. The study innovatively integrates the advantages of traditional Chinese medicine moxibustion for warming and promoting meridians and the low-intensity exercise of the modified Baduanjin, optimizes the difficulty of traditional rehabilitation training, and provides evidence-based basis for improving patient compliance and standardizing postoperative rehabilitation programs.

ELIGIBILITY:
Inclusion Criteria:

* ① Refer to the diagnostic criteria for LDH in the "Diagnosis and Treatment Guidelines for Lumbar Intervertebral Disc Protrusion (2020 Edition)";

  * Age > 18 years old; ③ Patients who have not responded to conservative treatment and have undergone minimally invasive surgery for lumbar intervertebral disc protrusion in our hospital, including percutaneous puncture interventional procedures (percutaneous intervertebral disc aspiration, percutaneous intervertebral disc laser ablation, percutaneous intervertebral disc ozone ablation, and radiofrequency nucleus removal and formation), micro-lumbar intervertebral disc resection, micro-endoscopic lumbar intervertebral disc resection, and percutaneous endoscopic lumbar intervertebral disc resection; ④ Participants who voluntarily participate in this study.

Exclusion Criteria:

* ① Previous history of lumbar surgery;

  * Those with severe spinal canal stenosis or other severe deformities;

    * Patients with bleeding tendencies or hematological diseases; ④ Patients with mental disorders and cognitive impairments; ⑤ Patients allergic to the drugs used in the study; ⑥ Patients with severe primary diseases (such as tuberculosis, tumors and mental disorders), or those with postoperative lumbar infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Japanese Orthopaedic Society,JOA | The 1st day after the operation, 1 month after the operation, 3 months after the operation
  JOA consists of three sections: daily life (0-14 points), subjective symptoms (0-9 points), and objective symptoms (0-6 points), with a total score of 29 points. The lower the score, the more obvious the functional impairment. The treatment improvement rate and efficacy are calculated based on the JOA score, using the formula: [(post-treatment score - pre-treatment score) ÷ (29 - pre-treatment score)] x 100%. Among them, an improvement rate of ≥ 75% is considered excellent; 50% - 74% is considered good; 25% - 49% is considered moderate improvement; 0% - 24% is considered poor. The efficacy judgment standard for the improvement rate is as follows: when the improvement rate is 100%, it is considered cured; when the improvement rate is greater than 60%, it is considered marked improvement; when it is 25% - 60%, it is considered effective; and when it is less than 25%, it is considered ineffective.

SECONDARY OUTCOMES:
Hamilton anxiety scale,HAMA | The 1st day after the operation, 1 month after the operation, 3 months after the operation
  This is used to assess the severity of anxiety symptoms. A total score of less than 7 indicates no anxiety symptoms; a score greater than 7 suggests the presence of anxiety; a score of 14 or above indicates the existence of anxiety; a score of 21 or above indicates significant anxiety; and a score of 29 or above may indicate severe anxiety.
Visual Analogue Scale，VAS | The 1st day after the operation, 1 month after the operation, 3 months after the operation
  Draw a 10-centimeter horizontal line on the paper. Mark one end of the line as 0cm, indicating no pain at all; mark the other end as 10cm, representing severe pain. Place the side with the scale facing away from the patient. Ask the patient to make a mark at the corresponding position on this line. The recorded scale value is the degree of pain the patient felt at that moment.

IPD SHARING:
Plan to Share IPD: Undecided